CLINICAL TRIAL: NCT03738475
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety, Pharmacodynamics, Efficacy, and Pharmacokinetics of TIMP-GLIA in Subjects With Well-controlled Celiac Disease Undergoing Oral Gluten Challenge
Brief Title: Study of the Safety, Pharmacodynamics, Efficacy, and PK of TIMP-GLIA in Subjects With Celiac Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: COUR Pharmaceutical Development Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TGLIA-5.002
Record Dates: First submitted 2018-11-09; First posted 2018-11-13 (Actual); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-07

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized double-blind placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TIMP-GLIA (Experimental): 8 mg/kg up to a maximum of 650 mg administered intravenously on days 1 and 8.
  Interventions: Drug: TIMP-GLIA
- Placebo (Placebo Comparator): Normal saline administered intravenously on days 1 and 8.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TIMP-GLIA — 8 mg/kg up to a maximum of 650 mg administered intravenously on days 1 and 8.
  Other Names: TAK-101
  Arms: TIMP-GLIA
Drug: Placebo — Administered intravenously on days 1 and 8.
  Other Names: 0.9% sodium chloride (normal saline)
  Arms: Placebo

SUMMARY:
Subjects enrolled in this study will be evaluated for immune responses and histological changes in the small bowel following 2 doses of TIMP-GLIA or placebo and a 14-day oral gluten challenge.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled clinical trial to assess the safety, pharmacodynamics, efficacy, and PK, of TIMP-GLIA in subjects with well-controlled celiac disease (CD) following an oral gluten challenge. Subjects aged 18 to 70 years inclusive, with documented history of biopsy-proven confirmed CD, and on a gluten-free diet (GFD) for a minimum of 6 months, will be screened. Subjects who meet all inclusion and no exclusion criteria, and provide written informed consent, will be randomized within 45 days after Screening to receive 2 intravenous (IV) infusions of TIMP-GLIA, 8 mg/kg up to a maximum of 650 mg or placebo (normal saline) in a 1:1 ratio. Treatment with drug or placebo will be followed by 14 days gluten challenge.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or nonpregnant female, ages 18 to 70 years inclusive, at Screening Visit.
2. Biopsy-confirmed CD (intestinal histology showing villous atrophy).
3. Positive for human leukocyte antigen (HLA)-DQ2 or HLA-DQ2/DQ8 - results will be obtained at Screening if unknown or results are not available.
4. Self-reported to be on a GFD for at least 6 months prior to Screening and agree to continue GFD throughout study, with the exception of the oral gluten challenge.

Normal or negative celiac serology, at screening, defined as:

1. Measurable total serum immunoglobulin A (IgA) AND
2. Negative or weak positive tissue transglutaminase (tTG) IgA titer OR
3. If IgA deficient, defined by a serum IgA level of < 3 mg/dL, negative or weak positive DGP- IgG titer.

   6. Vh:Cd ≥ 1.5 on screening biopsy.

   Key Exclusion Criteria:
   1. Positive for only HLA-DQ8.
   2. History of clinically confirmed immunoglobulin E (IgE)-mediated reaction and/or anaphylaxis to wheat (i.e., "wheat allergy"), barley or rye.
   3. Uncontrolled CD and/or active signs/symptoms of CD, in the opinion of the investigator.
   4. Untreated or active gastrointestinal disease such as peptic ulcer disease, esophagitis (Los Angeles Classification ≥ Grade C), irritable bowel syndrome, inflammatory bowel disease, or microscopic colitis.
   5. Immunocompromised individuals, including those receiving immunosuppressive doses of corticosteroids (more than 20 mg of prednisone given daily or on alternative days for 2 weeks or more within 6 months prior Dose 1, any dose of corticosteroids within 30 days of Day 1, or high dose inhaled corticosteroids [> 960 µg/day of beclomethasone dipropionate or equivalent]) or other immunosuppressive agents.
   6. Presence or history of celiac-associated thyroid disease or Type 1 diabetes, regardless of current treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (8):
- United States (8):
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Advanced Clinical Research, Meridian, Idaho
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Prism Clinical Research, Saint Paul, Minnesota
  - Rapid Medical Research, Beachwood, Ohio
  - Advanced Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Kelly CP, Murray JA, Leffler DA, Getts DR, Bledsoe AC, Smithson G, First MR, Morris A, Boyne M, Elhofy A, Wu TT, Podojil JR, Miller SD; TAK-101 Study Group. TAK-101 Nanoparticles Induce Gluten-Specific Tolerance in Celiac Disease: A Randomized, Double-Blind, Placebo-Controlled Study. Gastroenterology. 2021 Jul;161(1):66-80.e8. doi: 10.1053/j.gastro.2021.03.014. Epub 2021 Mar 17. PMID 33722583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in the United States from 11 November 2018 to 22 July 2019.
Pre-assignment Details: Participants diagnosed with celiac disease (CD) were enrolled in a 1:1 ratio in one of two treatment groups: Tolerogenic Immune Modifying Particles - Gliadin (TIMP-GLIA) or Placebo.
Groups:
- TIMP-GLIA 8 mg/kg: TIMP-GLIA 8 milligram per kilogram (mg/kg), infusion, intravenously, once on Days 1 and 8.
- Placebo: TIMP-GLIA placebo-matching infusion, intravenously, once on Days 1 and 8.
Period: Overall Study
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Started | 16 | 18
Completed | 15 | 18
Not Completed | 1 | 0
Not completed — Participant Non-Compliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all randomized participants who received at least one dose of study medication.
Groups:
- TIMP-GLIA 8 mg/kg: TIMP-GLIA 8 mg/kg, infusion, intravenously, once on Days 1 and 8.
- Total: Total of all reporting groups
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (13.47) | 42.2 (16.71) | 43.3 (15.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 18 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 18 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 18 | 34
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 28.213 (4.8479) | 27.100 (4.8214) | 27.624 (4.7933)
Disease Duration [Median (Full Range); unit: years] | 9.30 [2.5 to 21.1] | 8.45 [1.3 to 20.2] | 8.95 [1.3 to 21.1]
Gluten Free Diet Duration [Median (Full Range); unit: months] | 111.10 [28.3 to 253.6] | 113.45 [13.0 to 268.0] | 111.10 [13.0 to 268.0]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Interferon-Gamma Spot Forming Units (IFN-gamma SFUs) in a Gliadin-specific Enzyme-linked Immunospot (ELISpot) at Day 20
Description: The spots formed by interferon-gamma-secreting T-cells were counted with an automated ELISPOT analyzer. The average spot-forming units (SFU) per antigen was calculated. A response was considered positive when the average SFU in wells with a given peptide was at least twice that of the average SFU in the no-peptide control wells. Baseline (Day 15/Day 1) was defined as Day 15 (or Day 1 if enough blood was not available on Day 15). Peripheral blood mononuclear cell is PBMC.
Time Frame: Baseline (Day 15/Day 1), Day 20
Population: The pharmacodynamic population included all randomized participants who received two doses of study medication, completed at least the first 3 days of the gluten challenge (12 grams per day [g/day] for 3 days), and had pharmacodynamic results on Study Days 1, 15, and 20.
Measure: Mean (Standard Deviation); unit: SFUs/10^6 cells PBMC
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 13 | 16
SFUs/10^6 cells PBMC
  Baseline (Day 15/Day 1) | 3.08 (5.263) | 1.98 (3.184)
  Change at Day 20 | 2.01 (6.958) | 17.57 (25.283)
Statistical Analysis 1: Comparison: TIMP-GLIA 8 mg/kg vs Placebo; Test type: Superiority; p = 0.0056, Wilcoxon Rank Sum test — Based on Wilcoxon Rank Sum test for the change from baseline between treatment groups

2. Secondary Outcome: Change From Baseline in Gliadin-specific T Cell Proliferation by Enzyme-linked Immunosorbent Assay (ELISA) at Day 20
Description: Gliadin-specific T cell proliferation was determined by ELISA test. Baseline (Day 15/Day 1) was defined as Day 15 (or Day 1 if enough blood was not available on Day 15).
Time Frame: Baseline (Day 15/Day 1), Day 20
Population: The pharmacodynamic population included all randomized participants who received two doses of study medication, completed at least the first 3 days of the gluten challenge (12 g/day for 3 days), and had pharmacodynamic results on Study Days 1, 15, and 20. Participants evaluable for this measure at given time point were included for the assessment.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 13 | 16
picogram per milliliter (pg/mL)
  Baseline (Day 15/Day 1): number analyzed (Participants) | 13 | 15
  Baseline (Day 15/Day 1) | 0.87 (0.275) | 1.00 (0.178)
  Change at Day 20: number analyzed (Participants) | 13 | 15
  Change at Day 20 | 0.05 (0.284) | 0.00 (0.180)

3. Secondary Outcome: Change From Baseline in Gliadin-specific T Cell Cytokine Secretion by ELISA at Day 20
Description: Gliadin-specific T Cell cytokine secretion was determined by ELISA test. Gliadin-specific cytokine included interferon gamma (IFN-γ), interleukin (IL) 1-beta (1-β), IL-10, IL-12, IL-13, IL-2, IL-4, IL-6, IL-8, tumor necrosis factor alpha (TNF-α). Baseline (Day 15/Day 1) was defined as Day 15 (or Day 1 if enough blood was not available on Day 15). A negative change from baseline value was reported when the observed sample response was less than the observed background response.
Time Frame: Baseline (Day 15/Day 1), Day 20
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 13 | 16
pg/mL
  Baseline (Day 15/Day 1): IFN-γ | 1.44 (2.727) | 1.70 (4.251)
  Change at Day 20: IFN-γ: number analyzed (Participants) | 12 | 15
  Change at Day 20: IFN-γ | -0.43 (2.044) | -0.01 (2.149)
  Baseline (Day 15/Day 1): IL1-β | 1.24 (1.507) | 2.68 (4.548)
  Change at Day 20: IL1-β: number analyzed (Participants) | 12 | 16
  Change at Day 20: IL1-β | 0.00 (1.456) | -0.12 (5.946)
  Baseline (Day 15/Day 1): IL-10: number analyzed (Participants) | 12 | 15
  Baseline (Day 15/Day 1): IL-10 | 0.42 (0.688) | 0.80 (1.135)
  Change at Day 20 :IL-10: number analyzed (Participants) | 8 | 13
  Change at Day 20 :IL-10 | 0.53 (0.754) | -0.21 (1.302)
  Baseline (Day 15/Day 1): IL-12: number analyzed (Participants) | 12 | 12
  Baseline (Day 15/Day 1): IL-12 | 0.23 (0.727) | -0.03 (0.755)
  Change at Day 20: IL-12: number analyzed (Participants) | 11 | 11
  Change at Day 20: IL-12 | -0.01 (0.616) | 0.13 (0.548)
  Baseline (Day 15/Day 1): IL-13: number analyzed (Participants) | 13 | 13
  Baseline (Day 15/Day 1): IL-13 | 2.23 (2.831) | 0.94 (3.504)
  Change at Day 20: IL-13: number analyzed (Participants) | 7 | 9
  Change at Day 20: IL-13 | -2.06 (5.700) | 0.36 (1.655)
  Baseline (Day 15/Day 1): IL-2: number analyzed (Participants) | 12 | 14
  Baseline (Day 15/Day 1): IL-2 | 1.00 (1.117) | 1.29 (1.510)
  Change at Day 20: IL-2: number analyzed (Participants) | 7 | 11
  Change at Day 20: IL-2 | 0.27 (1.180) | 0.20 (0.932)
  Baseline (Day 15/Day 1): IL-4: number analyzed (Participants) | 13 | 15
  Baseline (Day 15/Day 1): IL-4 | 0.12 (0.180) | 0.19 (0.388)
  Change at Day 20: IL-4: number analyzed (Participants) | 10 | 13
  Change at Day 20: IL-4 | -0.07 (0.227) | -0.09 (0.434)
  Baseline (Day 15/Day 1): IL-6: number analyzed (Participants) | 13 | 15
  Baseline (Day 15/Day 1): IL-6 | -0.59 (18.704) | 32.06 (123.405)
  Change at Day 20: IL-6: number analyzed (Participants) | 12 | 15
  Change at Day 20: IL-6 | 12.76 (29.303) | -16.88 (131.535)
  Baseline (Day 15/Day 1): IL-8: number analyzed (Participants) | 12 | 14
  Baseline (Day 15/Day 1): IL-8 | 0.03 (0.091) | 0.00 (0.007)
  Change at Day 20: IL-8: number analyzed (Participants) | 12 | 14
  Change at Day 20: IL-8 | -0.03 (0.091) | 0.00 (0.007)
  Baseline (Day 15/Day 1): TNF-α: number analyzed (Participants) | 13 | 15
  Baseline (Day 15/Day 1): TNF-α | 2.25 (2.763) | 11.75 (27.434)
  Change at Day 20: TNF-α: number analyzed (Participants) | 9 | 13
  Change at Day 20: TNF-α | 3.20 (3.099) | -1.95 (33.181)

4. Secondary Outcome: Change From Baseline in Gut-Homing CD4, CD8 and Gamma Delta T-cells by Mass Cytometry (CyTOF) at Day 20
Description: Change from baseline value for Gut-Homing cells like CD4, CD8 and Gamma Delta T-cells were reported. Baseline (Day 15/Day 1) was defined as Day 15 (or Day 1 if enough blood was not available on Day 15). Phenotype (unique cell population) for CD8 cell is EM CD8 > aE+b7hi > aE+b7hiCD38+, for CD4 is EM Th > a4+b7hi > a4+b7hiCD38+ and for Gamma Delta T-cells is TCRgd T cells > aE+b7hi > aE+b7hiCD38+ in this outcome measure.
Time Frame: Baseline (Day 15/Day 1), Day 20
Population: The pharmacodynamic population included all randomized participants who received two doses of study medication, completed at least the first 3 days of the gluten challenge (12 g/day for 3 days), and had pharmacodynamic results on Study Days 1, 15, and 20.
Measure: Mean (Standard Deviation); unit: percent parent
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 13 | 16
percent parent
  Baseline (Day 15/Day 1): CD8 | 0.21 (0.216) | 0.18 (0.285)
  Change at Day 20: CD8 | 0.69 (0.979) | 3.64 (3.685)
  Baseline (Day 15/Day 1): CD4 | 0.19 (0.210) | 0.16 (0.189)
  Change at Day 20: CD4 | 0.26 (0.549) | 1.05 (1.223)
  Baseline (Day 15/Day 1): Gamma Delta T-cells | 0.20 (0.186) | 0.13 (0.318)
  Change at Day 20: Gamma Delta T-cells | 0.15 (0.378) | 1.59 (2.598)

5. Secondary Outcome: Change From Baseline in Ratio of Villus Height to Crypt Depth (Vh:Cd) at Day 29
Description: Attenuation of the effects of gluten exposure was assessed by measuring the change from baseline in villous height (Vh) to crypt depth (Cd) ratio after 29 days of gluten challenge. Villi were the small finger like projections that line the small intestine and promote nutrient absorption and are often shortened in participants with CD. Crypts are grooves between the villi that are often elongated in participants with CD. A decreased Vh:Cd ratio indicates worsening disease. Baseline was defined as the last sample collected prior to the first dose of study medication (Screening Period) on Day 1.
Time Frame: Baseline (Screening), Day 29
Population: The histology population included all randomized participants who received two doses of study medication, completed the gluten challenge per protocol, and had both a baseline and Day 29 biopsy.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 13 | 15
ratio
  Baseline (Screening): Vh:Cd | 2.82 (0.306) | 3.01 (0.451)
  Change at Day 29: Vh:Cd: | -0.18 (0.381) | -0.63 (0.657)
Statistical Analysis 1: Comparison: TIMP-GLIA 8 mg/kg vs Placebo; Test type: Superiority; p = 0.0799, Wilcoxon Rank Sum test — Based on Wilcoxon Rank Sum test for the change from baseline between treatment groups

6. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (>=) 0.4 Decrease in Vh:Cd at Day 29
Description: Villi were the small finger like projections that line the small intestine and promote nutrient absorption and are often shortened in participants with CD. Crypts are grooves between the villi that are often elongated in participants with CD. A decreased Vh:Cd ratio indicates worsening disease.
Time Frame: Day 29
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 13 | 15
percentage of participants | 23.1 | 53.3

7. Secondary Outcome: Change From Baseline in Number of Intestinal Intraepithelial Lymphocytes (IELs) at Day 29
Description: IELs were white blood cells interspersed between epithelial cells of the small and large intestine where they function to preserve the integrity of the mucosal barrier by protecting the epithelium against pathogen or immune-induced pathology. Increased intraepithelial lymphocytes was associated with celiac disease. Baseline was defined as the last sample collected prior to the first dose of study medication (Screening Period) on Day 1.
Time Frame: Baseline (Screening), Day 29
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cells per 100 enterocytes
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 13 | 15
cells per 100 enterocytes
  Baseline (Screening): IELs | 39.62 (18.842) | 34.53 (12.389)
  Change at Day 29: IELs | 28.62 (19.241) | 35.00 (18.756)
Statistical Analysis 1: Comparison: TIMP-GLIA 8 mg/kg vs Placebo; Test type: Superiority; p = 0.2890, Wilcoxon Rank Sum test — Based on Wilcoxon Rank Sum test for the change from baseline between treatment groups

8. Secondary Outcome: Number of Participants Based on Celiac Symptom Index-Modified (CSI-M) Questionnaire Results by Treatment
Description: The CSI were clinically oriented, easily administered, questionnaires with 16 items. The modified CSI (6-items) was derived from a subset of questions from the CSI questionnaire, including the diarrhea, nausea, rumbling in stomach, stomach felt bloated, diarrhea and low energy level abdominal pain domains (a total of 6 questions), which were each assessed on a scale of 1 to 5- none of the time, a little of the time, some of the time, most of the time and all of the time respectively. Higher CSI scores correlate with more severe CD symptoms. It is to be used to assess symptoms before, during, and after the oral gluten challenge. Here D refers to Day.
Time Frame: Days 15, 20, 29 and 35
Population: The safety population included all randomized participants who received at least one dose of study medication. Here, "number analyzed" signifies the participants who were evaluable for this outcome measure for given time points.
Measure: Number; unit: participants
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 16 | 18
participants
  D 15, Pain/discomfort in abdomen/stomach: None | 11 | 13
  D 15, Pain/discomfort in abdomen/stomach: A little | 3 | 4
  D 15, Pain/discomfort in abdomen/stomach: Some | 2 | 1
  D 15, Pain/discomfort in abdomen/stomach: Most | 0 | 0
  D 15, Pain/discomfort in abdomen/stomach: All time | 0 | 0
  D 15, Nausea: None | 12 | 15
  D 15, Nausea: A little | 2 | 2
  D 15, Nausea: Some | 1 | 1
  D 15, Nausea: Most | 1 | 0
  D 15, Nausea: All time | 0 | 0
  D 15, Rumbling in stomach: None | 12 | 11
  D 15, Rumbling in stomach: A little | 2 | 5
  D 15, Rumbling in stomach: Some | 2 | 2
  D 15, Rumbling in stomach: Most | 0 | 0
  D 15, Rumbling in stomach: All time | 0 | 0
  D 15, Stomach felt bloated: None | 11 | 10
  D 15, Stomach felt bloated: A little | 4 | 7
  D 15, Stomach felt bloated: Some | 1 | 0
  D 15, Stomach felt bloated: Most | 0 | 1
  D 15, Stomach felt bloated: All time | 0 | 0
  D 15, Diarrhea: None | 14 | 15
  D 15, Diarrhea: A little | 2 | 3
  D 15, Diarrhea: Some | 0 | 0
  D 15, Diarrhea: Most | 0 | 0
  D 15, Diarrhea: All time | 0 | 0
  D 15, Low energy level: None | 6 | 11
  D 15, Low energy level: A little | 5 | 5
  D 15, Low energy level: Some | 3 | 1
  D 15, Low energy level: Most | 2 | 1
  D 15, Low energy level: All time | 0 | 0
  D 20, Pain/discomfort in abdomen/stomach: None: number analyzed (Participants) | 14 | 18
  D 20, Pain/discomfort in abdomen/stomach: None | 5 | 8
  D 20, Pain/discomfort in abdomen/stomach: A little: number analyzed (Participants) | 14 | 18
  D 20, Pain/discomfort in abdomen/stomach: A little | 4 | 3
  D 20, Pain/discomfort in abdomen/stomach: Some: number analyzed (Participants) | 14 | 18
  D 20, Pain/discomfort in abdomen/stomach: Some | 2 | 4
  D 20, Pain/discomfort in abdomen/stomach: Most: number analyzed (Participants) | 14 | 18
  D 20, Pain/discomfort in abdomen/stomach: Most | 3 | 2
  D 20, Pain/discomfort in abdomen/stomach: All time: number analyzed (Participants) | 14 | 18
  D 20, Pain/discomfort in abdomen/stomach: All time | 0 | 1
  D 20, Nausea: None: number analyzed (Participants) | 14 | 18
  D 20, Nausea: None | 4 | 5
  D 20, Nausea: A little: number analyzed (Participants) | 14 | 18
  D 20, Nausea: A little | 5 | 7
  D 20, Nausea: Some: number analyzed (Participants) | 14 | 18
  D 20, Nausea: Some | 3 | 3
  D 20, Nausea: Most: number analyzed (Participants) | 14 | 18
  D 20, Nausea: Most | 1 | 2
  D 20, Nausea: All time: number analyzed (Participants) | 14 | 18
  D 20, Nausea: All time | 1 | 1
  D 20, Rumbling in stomach: None: number analyzed (Participants) | 14 | 18
  D 20, Rumbling in stomach: None | 6 | 6
  D 20, Rumbling in stomach: A little: number analyzed (Participants) | 14 | 18
  D 20, Rumbling in stomach: A little | 2 | 6
  D 20, Rumbling in stomach: Some: number analyzed (Participants) | 14 | 18
  D 20, Rumbling in stomach: Some | 4 | 3
  D 20, Rumbling in stomach: Most: number analyzed (Participants) | 14 | 18
  D 20, Rumbling in stomach: Most | 1 | 2
  D 20, Rumbling in stomach: All time: number analyzed (Participants) | 14 | 18
  D 20, Rumbling in stomach: All time | 1 | 1
  D 20, Stomach felt bloated: None: number analyzed (Participants) | 14 | 18
  D 20, Stomach felt bloated: None | 7 | 4
  D 20, Stomach felt bloated: A little: number analyzed (Participants) | 14 | 18
  D 20, Stomach felt bloated: A little | 2 | 8
  D 20, Stomach felt bloated: Some: number analyzed (Participants) | 14 | 18
  D 20, Stomach felt bloated: Some | 1 | 3
  D 20, Stomach felt bloated: Most: number analyzed (Participants) | 14 | 18
  D 20, Stomach felt bloated: Most | 2 | 1
  D 20, Stomach felt bloated: All time: number analyzed (Participants) | 14 | 18
  D 20, Stomach felt bloated: All time | 2 | 2
  D 20, Diarrhea: None: number analyzed (Participants) | 14 | 18
  D 20, Diarrhea: None | 8 | 11
  D 20, Diarrhea: A little: number analyzed (Participants) | 14 | 18
  D 20, Diarrhea: A little | 2 | 4
  D 20, Diarrhea: Some: number analyzed (Participants) | 14 | 18
  D 20, Diarrhea: Some | 3 | 3
  D 20, Diarrhea: Most: number analyzed (Participants) | 14 | 18
  D 20, Diarrhea: Most | 1 | 0
  D 20, Diarrhea: All time: number analyzed (Participants) | 14 | 18
  D 20, Diarrhea: All time | 0 | 0
  D 20, Low energy level: None: number analyzed (Participants) | 14 | 18
  D 20, Low energy level: None | 3 | 6
  D 20, Low energy level: A little: number analyzed (Participants) | 14 | 18
  D 20, Low energy level: A little | 5 | 6
  D 20, Low energy level: Some: number analyzed (Participants) | 14 | 18
  D 20, Low energy level: Some | 0 | 2
  D 20, Low energy level: Most: number analyzed (Participants) | 14 | 18
  D 20, Low energy level: Most | 4 | 2
  D 20, Low energy level: All time: number analyzed (Participants) | 14 | 18
  D 20, Low energy level: All time | 2 | 2
  D 29, Pain/discomfort in abdomen/stomach: None: number analyzed (Participants) | 13 | 18
  D 29, Pain/discomfort in abdomen/stomach: None | 6 | 10
  D 29, Pain/discomfort in abdomen/stomach: A little: number analyzed (Participants) | 13 | 18
  D 29, Pain/discomfort in abdomen/stomach: A little | 2 | 5
  D 29, Pain/discomfort in abdomen/stomach: Some: number analyzed (Participants) | 13 | 18
  D 29, Pain/discomfort in abdomen/stomach: Some | 4 | 2
  D 29, Pain/discomfort in abdomen/stomach: Most: number analyzed (Participants) | 13 | 18
  D 29, Pain/discomfort in abdomen/stomach: Most | 1 | 0
  D 29, Pain/discomfort in abdomen/stomach: All time: number analyzed (Participants) | 13 | 18
  D 29, Pain/discomfort in abdomen/stomach: All time | 0 | 1
  D 29, Nausea: None: number analyzed (Participants) | 13 | 18
  D 29, Nausea: None | 8 | 9
  D 29, Nausea: A little: number analyzed (Participants) | 13 | 18
  D 29, Nausea: A little | 3 | 5
  D 29, Nausea: Some: number analyzed (Participants) | 13 | 18
  D 29, Nausea: Some | 1 | 1
  D 29, Nausea: Most: number analyzed (Participants) | 13 | 18
  D 29, Nausea: Most | 1 | 2
  D 29, Nausea: All time: number analyzed (Participants) | 13 | 18
  D 29, Nausea: All time | 0 | 1
  D 29, Rumbling in stomach: None: number analyzed (Participants) | 13 | 18
  D 29, Rumbling in stomach: None | 7 | 9
  D 29, Rumbling in stomach: A little: number analyzed (Participants) | 13 | 18
  D 29, Rumbling in stomach: A little | 1 | 5
  D 29, Rumbling in stomach: Some: number analyzed (Participants) | 13 | 18
  D 29, Rumbling in stomach: Some | 3 | 2
  D 29, Rumbling in stomach: Most: number analyzed (Participants) | 13 | 18
  D 29, Rumbling in stomach: Most | 2 | 1
  D 29, Rumbling in stomach: All time: number analyzed (Participants) | 13 | 18
  D 29, Rumbling in stomach: All time | 0 | 1
  D 29, Stomach felt bloated: None: number analyzed (Participants) | 13 | 18
  D 29, Stomach felt bloated: None | 7 | 8
  D 29, Stomach felt bloated: A little: number analyzed (Participants) | 13 | 18
  D 29, Stomach felt bloated: A little | 1 | 6
  D 29, Stomach felt bloated: Some: number analyzed (Participants) | 13 | 18
  D 29, Stomach felt bloated: Some | 2 | 1
  D 29, Stomach felt bloated: Most: number analyzed (Participants) | 13 | 18
  D 29, Stomach felt bloated: Most | 2 | 2
  D 29, Stomach felt bloated: All time: number analyzed (Participants) | 13 | 18
  D 29, Stomach felt bloated: All time | 1 | 1
  D 29, Diarrhea: None: number analyzed (Participants) | 13 | 18
  D 29, Diarrhea: None | 10 | 13
  D 29, Diarrhea: A little: number analyzed (Participants) | 13 | 18
  D 29, Diarrhea: A little | 1 | 3
  D 29, Diarrhea: Some: number analyzed (Participants) | 13 | 18
  D 29, Diarrhea: Some | 2 | 1
  D 29, Diarrhea: Most: number analyzed (Participants) | 13 | 18
  D 29, Diarrhea: Most | 0 | 0
  D 29, Diarrhea: All time: number analyzed (Participants) | 13 | 18
  D 29, Diarrhea: All time | 0 | 1
  D 29, Low energy level: None: number analyzed (Participants) | 13 | 18
  D 29, Low energy level: None | 4 | 8
  D 29, Low energy level: A little: number analyzed (Participants) | 13 | 18
  D 29, Low energy level: A little | 3 | 6
  D 29, Low energy level: Some: number analyzed (Participants) | 13 | 18
  D 29, Low energy level: Some | 2 | 3
  D 29, Low energy level: Most: number analyzed (Participants) | 13 | 18
  D 29, Low energy level: Most | 3 | 0
  D 29, Low energy level: All time: number analyzed (Participants) | 13 | 18
  D 29, Low energy level: All time | 1 | 1
  D 35, Pain/discomfort in abdomen/stomach: None: number analyzed (Participants) | 13 | 18
  D 35, Pain/discomfort in abdomen/stomach: None | 8 | 15
  D 35, Pain/discomfort in abdomen/stomach: A little: number analyzed (Participants) | 13 | 18
  D 35, Pain/discomfort in abdomen/stomach: A little | 4 | 2
  D 35, Pain/discomfort in abdomen/stomach: Some: number analyzed (Participants) | 13 | 18
  D 35, Pain/discomfort in abdomen/stomach: Some | 1 | 1
  D 35, Pain/discomfort in abdomen/stomach: Most: number analyzed (Participants) | 13 | 18
  D 35, Pain/discomfort in abdomen/stomach: Most | 0 | 0
  D 35, Pain/discomfort in abdomen/stomach: All time: number analyzed (Participants) | 13 | 18
  D 35, Pain/discomfort in abdomen/stomach: All time | 0 | 0
  D 35, Nausea: None: number analyzed (Participants) | 13 | 18
  D 35, Nausea: None | 9 | 16
  D 35, Nausea: A little: number analyzed (Participants) | 13 | 18
  D 35, Nausea: A little | 2 | 2
  D 35, Nausea: Some: number analyzed (Participants) | 13 | 18
  D 35, Nausea: Some | 2 | 0
  D 35, Nausea: Most: number analyzed (Participants) | 13 | 18
  D 35, Nausea: Most | 0 | 0
  D 35, Nausea: All time: number analyzed (Participants) | 13 | 18
  D 35, Nausea: All time | 0 | 0
  D 35, Rumbling in stomach: None: number analyzed (Participants) | 13 | 18
  D 35, Rumbling in stomach: None | 10 | 11
  D 35, Rumbling in stomach: A little: number analyzed (Participants) | 13 | 18
  D 35, Rumbling in stomach: A little | 1 | 7
  D 35, Rumbling in stomach: Some: number analyzed (Participants) | 13 | 18
  D 35, Rumbling in stomach: Some | 2 | 0
  D 35, Rumbling in stomach: Most: number analyzed (Participants) | 13 | 18
  D 35, Rumbling in stomach: Most | 0 | 0
  D 35, Rumbling in stomach: All time: number analyzed (Participants) | 13 | 18
  D 35, Rumbling in stomach: All time | 0 | 0
  D 35, Stomach felt bloated: None: number analyzed (Participants) | 13 | 18
  D 35, Stomach felt bloated: None | 8 | 10
  D 35, Stomach felt bloated: A little: number analyzed (Participants) | 13 | 18
  D 35, Stomach felt bloated: A little | 3 | 6
  D 35, Stomach felt bloated: Some: number analyzed (Participants) | 13 | 18
  D 35, Stomach felt bloated: Some | 2 | 2
  D 35, Stomach felt bloated: Most: number analyzed (Participants) | 13 | 18
  D 35, Stomach felt bloated: Most | 0 | 0
  D 35, Stomach felt bloated: All time: number analyzed (Participants) | 13 | 18
  D 35, Stomach felt bloated: All time | 0 | 0
  D 35, Diarrhea: None: number analyzed (Participants) | 13 | 18
  D 35, Diarrhea: None | 11 | 14
  D 35, Diarrhea: A little: number analyzed (Participants) | 13 | 18
  D 35, Diarrhea: A little | 2 | 3
  D 35, Diarrhea: Some: number analyzed (Participants) | 13 | 18
  D 35, Diarrhea: Some | 0 | 0
  D 35, Diarrhea: Most: number analyzed (Participants) | 13 | 18
  D 35, Diarrhea: Most | 0 | 1
  D 35, Diarrhea: All time: number analyzed (Participants) | 13 | 18
  D 35, Diarrhea: All time | 0 | 0
  D 35, Low energy level: None: number analyzed (Participants) | 13 | 18
  D 35, Low energy level: None | 7 | 14
  D 35, Low energy level: A little: number analyzed (Participants) | 13 | 18
  D 35, Low energy level: A little | 1 | 2
  D 35, Low energy level: Some: number analyzed (Participants) | 13 | 18
  D 35, Low energy level: Some | 4 | 0
  D 35, Low energy level: Most: number analyzed (Participants) | 13 | 18
  D 35, Low energy level: Most | 1 | 2
  D 35, Low energy level: All time: number analyzed (Participants) | 13 | 18
  D 35, Low energy level: All time | 0 | 0

9. Secondary Outcome: Plasma Concentrations of TIMP-GLIA
Time Frame: Day 8: 0 hours (pre-infusion), end of infusion, and at 2 hours post-infusion
Population: The pharmacokinetic population included all randomized participants who received two doses of study medication and had at least one reported concentration. The pharmacokinetic population where data at specified time points were available.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | TIMP-GLIA 8 mg/kg
Number analyzed (Participants) | 16
nanogram per milliliter (ng/mL)
  0 hours (pre-infusion) | 13.06 (52.250)
  End of Infusion | 684.54 (319.069)
  2 hours post infusion: number analyzed (Participants) | 15
  2 hours post infusion | 383.46 (153.225)

10. Secondary Outcome: Number of Participants Who Experience at Least 1 Treatment-emergent Adverse Event (TEAE) and Serious Adverse Event (SAE)
Time Frame: From the first dose of study drug up to Day 35
Population: The safety population included all randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 16 | 18
Participants
  TEAE | 16 | 18
  SAE | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Time Frame: From the first dose of study drug up to Day 35
Population: The safety population included all randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 16 | 18
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Hematology or Serum Chemistry Laboratory Values
Time Frame: From the first dose of study drug up to Day 35
Population: The safety population included all randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 16 | 18
Participants | 0 | 0

13. Secondary Outcome: Change From Baseline in Deamidated Gliadin Peptide Immunoglobulin G (DGP-IgG) Antibodies at Days 8, 15, 20, 29, and 35
Description: Baseline was defined as the last sample collected prior to the first dose of study medication (Screening Period) on Day 1.
Time Frame: Baseline (Screening), Days 8, 15, 20, 29, and 35
Population: The safety population included all randomized participants who received at least one dose of study medication. Participants evaluable for this measure at given time point were included for the assessment.
Measure: Mean (Standard Deviation); unit: units
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 16 | 18
units
  Baseline (Screening) | 7.9 (11.53) | 5.9 (3.48)
  Change at Day 8 | 4.3 (7.43) | -0.6 (1.58)
  Change at Day 15 | 27.8 (28.92) | 0.3 (1.67)
  Change at Day 20: number analyzed (Participants) | 14 | 17
  Change at Day 20 | 28.6 (29.63) | -0.1 (1.76)
  Change at Day 29: number analyzed (Participants) | 13 | 18
  Change at Day 29 | 28.4 (31.27) | 8.9 (13.23)
  Change at Day 35: number analyzed (Participants) | 13 | 18
  Change at Day 35 | 28.4 (29.68) | 20.7 (27.04)

14. Secondary Outcome: Change From Baseline in Serum Complement Levels of C3a and SC5B-9 at Days 2, 8, 9, and 15
Description: Baseline was defined as the pre-dose value on Day 1.
Time Frame: Baseline (Day 1), Days 2, 8, 9, and 15
Population: The safety population included all randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 16 | 18
ng/mL
  Baseline (Day 1): C3a | 1024.0 (430.15) | 1069.9 (435.78)
  Change at Day 2: C3a | -144.6 (452.51) | 112.3 (1086.95)
  Change at Day 8: C3a | 244.7 (449.20) | -115.3 (385.44)
  Change at Day 9: C3a | -63.0 (227.28) | -71.2 (441.80)
  Change at Day 15: C3a | -165.2 (308.01) | 54.8 (603.56)
  Baseline (Day 1): SC5B-9 | 130.5 (44.69) | 114.7 (40.68)
  Change at Day 2: SC5B-9 | -8.7 (25.83) | -4.5 (20.18)
  Change at Day 8: SC5B-9 | 866.5 (924.08) | -4.6 (28.72)
  Change at Day 9: SC5B-9 | 40.5 (137.83) | -4.8 (37.18)
  Change at Day 15: SC5B-9 | 5.5 (57.06) | 18.4 (53.46)

15. Secondary Outcome: Change From Baseline in Serum Complement Levels of C5a at Days 2, 8, 9, and 15
Description: Baseline was defined as the pre-dose value on Day 1.
Time Frame: Baseline (Day 1) , Days 2, 8, 9, and 15
Population: The safety population included all randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 16 | 18
microgram per liter (mcg/L)
  Baseline (Day 1) | 9.290 (6.5091) | 7.267 (3.2526)
  Change at Day 2 | 0.763 (1.0587) | -0.067 (0.6776)
  Change at Day 8 | 8.373 (8.0077) | 0.082 (0.7604)
  Change at Day 9 | 0.926 (1.3873) | 0.347 (1.0356)
  Change at Day 15 | 0.319 (1.7868) | 0.241 (0.9151)

16. Secondary Outcome: Change From Baseline in Serum Complement Levels of C1q Binding at Days 15, 20, 29, and 35
Description: Baseline was defined as the pre-dose value on Day 1.
Time Frame: Baseline (Day 1), Days 15, 20, 29, and 35
Population: The safety population included all randomized participants who received at least one dose of study medication. Participants who were evaluable for this measure at given time point were included for the assessment.
Measure: Mean (Standard Deviation); unit: units per milliliter (U/mL)
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 16 | 18
units per milliliter (U/mL)
  Baseline (Day 1) | 3.65 (2.026) | 4.53 (1.962)
  Change at Day 15 | 0.64 (1.249) | 0.21 (1.498)
  Change at Day 20: number analyzed (Participants) | 13 | 18
  Change at Day 20 | 0.88 (1.315) | -0.15 (1.274)
  Change at Day 29: number analyzed (Participants) | 13 | 18
  Change at Day 29 | 0.10 (1.901) | 0.18 (2.073)
  Change at Day 35: number analyzed (Participants) | 13 | 18
  Change at Day 35 | 0.49 (1.310) | 0.09 (2.116)

17. Secondary Outcome: Change From Baseline in Serum Cytokines (IFN-γ, IL 1-β, IL-2, IL-4, IL-6, IL-8 , IL-10, IL-12p70, and TNF-Alpha) at Days 2, 8, 9, and 15
Description: Baseline was defined as Day 1 pre-dose. A negative change from baseline value was reported when the observed sample response was less than the observed background response.
Time Frame: Baseline (Day 1), Days 2, 8, 9, and 15
Population: The safety population included all randomized participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
Number analyzed (Participants) | 16 | 18
pg/mL
  Baseline (Day 1): IFN-γ | 7.375 (9.5787) | 4.592 (1.9801)
  Change at Day 2: IFN-γ | 9.871 (19.3167) | -0.179 (0.8403)
  Change at Day 8: IFN-γ | -2.374 (10.3311) | 5.245 (15.7119)
  Change at Day 9: IFN-γ | 1.663 (14.7044) | 3.709 (12.0744)
  Change at Day 15: IFN-γ | 0.539 (12.8988) | 0.871 (2.4732)
  Baseline (Day 1): IL1-β | 0.600 (0.0000) | 0.600 (0.0000)
  Change at Day 2: IL1-β | 0.000 (0.0000) | 0.0000 (0.0000)
  Change at Day 8: IL1-β | 0.000 (0.000) | 0.0000 (0.0000)
  Change at Day 9: IL1-β | 0.000 (0.000) | 0.0000 (0.0000)
  Change at Day 15: IL1-β | 0.000 (0.000) | 0.0000 (0.0000)
  Baseline (Day 1): IL-2 | 0.731 (0.0450) | 0.824 (0.4431)
  Change at Day 2: IL-2 | 0.004 (0.0175) | 0.001 (0.0047)
  Change at Day 8: IL-2 | 0.008 (0.0325) | -0.021 (0.0872)
  Change at Day 9: IL-2 | 0.006 (0.0250) | -0.022 (0.0943)
  Change at Day 15: IL-2 | 0.006 (0.0250) | -0.023 (0.0990)
  Baseline (Day 1): IL-4 | 0.380 (0.0000) | 0.380 (0.0000)
  Change at Day 2: IL-4 | 0.000 (0.000) | 0.0000 (0.0000)
  Change at Day 8: IL-4 | 0.000 (0.000) | 0.0000 (0.0000)
  Change at Day 9: IL-4 | 0.000 (0.000) | 0.0000 (0.0000)
  Change at Day 15: IL-4 | 0.000 (0.000) | 0.0000 (0.0000)
  Baseline (Day 1): IL-6 | 1.067 (0.3473) | 1.005 (0.1621)
  Change at Day 2: IL-6 | -0.009 (0.0924) | 0.069 (0.2733)
  Change at Day 8: IL-6 | 0.024 (0.3507) | 0.169 (0.6991)
  Change at Day 9: IL-6 | 0.159 (0.4817) | 0.051 (0.2330)
  Change at Day 15: IL-6 | -0.059 (0.3768) | -0.008 (0.1400)
  Baseline (Day 1): IL-8 | 12.602 (5.7067) | 11.497 (3.9699)
  Change at Day 2: IL-8 | 11.159 (17.5276) | 0.236 (5.6791)
  Change at Day 8: IL-8 | -0.470 (3.1986) | -2.177 (3.1075)
  Change at Day 9: IL-8 | 5.816 (9.5328) | -1.685 (4.1328)
  Change at Day 15: IL-8 | -1.959 (5.0839) | -1.394 (4.0435)
  Baseline (Day 1): IL-10 | 1.784 (5.4054) | 0.449 (0.1651)
  Change at Day 2: IL-10 | 0.081 (0.0969) | 0.042 (0.1403)
  Change at Day 8: IL-10 | -0.040 (0.2209) | 0.017 (0.1701)
  Change at Day 9: IL-10 | 0.494 (1.2476) | 0.067 (0.1695)
  Change at Day 15: IL-10 | 0.307 (1.0885) | -0.013 (0.0531)
  Baseline (Day 1): IL-12p70 | 3.280 (0.0000) | 3.280 (0.0000)
  Change at Day 2: IL-12p70 | 0.0000 (0.0000) | 0.0000 (0.0000)
  Change at Day 8: IL-12p70 | 0.0000 (0.0000) | 0.0000 (0.0000)
  Change at Day 9: IL-12p70 | 0.0000 (0.0000) | 0.0000 (0.0000)
  Change at Day 15: IL-12p70 | 0.0000 (0.0000) | 0.0000 (0.0000)
  Baseline (Day 1): TNF-α | 2.856 (0.6101) | 2.421 (0.6177)
  Change at Day 2: TNF-α | 1.218 (1.1446) | -0.037 (0.4394)
  Change at Day 8: TNF-α | 0.132 (0.5762) | 0.080 (0.3451)
  Change at Day 9: TNF-α | 0.801 (0.7369) | -0.043 (0.3940)
  Change at Day 15: TNF-α | 0.138 (0.7129) | 0.083 (0.2492)

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events that started after the first dose of study drug up to Day 35
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TIMP-GLIA 8 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 16/16 | 18/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIMP-GLIA 8 mg/kg (N=16) | Placebo (N=18)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 5
Abdominal distension (Gastrointestinal disorders) | 9 | 11
Abdominal pain (Gastrointestinal disorders) | 6 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 9
Erosive duodenitis (Gastrointestinal disorders) | 0 | 1
Eructation (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 6 | 7
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 13 | 13
Oesophageal mucosa erythema (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 5 | 6
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 3 | 0
Chest discomfort (General disorders) | 2 | 0
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 5 | 9
Feeling abnormal (General disorders) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Urinary bladder abscess (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 3
Head discomfort (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 7 | 3
Lethargy (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 2 | 0
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT03738475/SAP_000.pdf
  • Study Protocol (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT03738475/Prot_001.pdf